CLINICAL TRIAL: NCT01304329
Title: Relative Bioavailability of BI 10773 and Simvastatin After Single and Combined Administration - an Open-label, Randomised, Crossover Trial in Healthy Subjects
Brief Title: Drug-drug Interaction of Empagliflozin (BI 10773) and Simvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.63; 2010-023680-18 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-02-21; First posted 2011-02-25 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Simvastatin

ARMS (3):
- treatment A, reference (Experimental): 1 tablet BI 10773, oral administration with 240 ml water
  Interventions: Drug: BI 10773
- treatment B, reference (Experimental): 1 tablet simvastatin, oral administration with 240 ml water
  Interventions: Drug: simvastatin
- treatment C, test (Experimental): 1 tablet BI 10773 + 1 tablet simvastatin, oral administration with 240 ml water
  Interventions: Drug: BI 10773; Drug: simvastatin

INTERVENTIONS:
Drug: BI 10773 — Medium dose oral administration
  Arms: treatment C, test
Drug: simvastatin — Medium dose oral administration
  Arms: treatment C, test
Drug: simvastatin — Medium dose oral administration
  Arms: treatment B, reference
Drug: BI 10773 — Medium dose oral administration
  Arms: treatment A, reference

SUMMARY:
The objective of the study is to investigate the drug-drug interaction potential between BI 10773 and simvastatin.

ELIGIBILITY:
Inclusion criteria:

- healthy male and female subjects

Exclusion criteria:

- Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.63.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, open label, 3 period crossover study. Treatment periods were separated by a washout period of at least 7 days.
Groups:
- Empa Alone / Simvastatin Alone / Empa Plus Sim: Patients were administered three treatments in the following order:
  * A single dose of empagliflozin 25mg
  * A single dose of simvastatin 40mg
  * A single dose of empagliflozin 25mg together with 40mg simvastatin
- Empa Alone / Empa Plus Sim / Simvastatin Alone: Patients were administered three treatments in the following order:
  * A single dose of empagliflozin 25mg
  * A single dose of empagliflozin 25mg together with 40mg simvastatin
  * A single dose of simvastatin 40mg
- Simvastatin Alone / Empa Alone / Empa Plus Sim: Patients were administered three treatments in the following order:
  * A single dose of simvastatin 40mg
  * A single dose of empagliflozin 25mg
  * A single dose of empagliflozin 25mg together with 40mg simvastatin
- Simvastatin Alone / Empa Plus Sim / Empa Alone: Patients were administered three treatments in the following order:
  * A single dose of simvastatin 40mg
  * A single dose of empagliflozin 25mg together with 40mg simvastatin
  * A single dose of empagliflozin 25mg
- Empa Plus Sim / Empa Alone / Simvastatin Alone: Patients were administered three treatments in the following order:
  * A single dose of empagliflozin 25mg together with 40mg simvastatin
  * A single dose of empagliflozin 25mg
  * A single dose of simvastatin 40mg
- Empa Plus Sim / Simvastatin Alone / Empa Alone: Patients were administered three treatments in the following order:
  * A single dose of empagliflozin 25mg together with 40mg simvastatin
  * A single dose of simvastatin 40mg
  * A single dose of empagliflozin 25mg
Period: First Intervention (3 Days)
Arm/Group | Empa Alone / Simvastatin Alone / Empa Plus Sim | Empa Alone / Empa Plus Sim / Simvastatin Alone | Simvastatin Alone / Empa Alone / Empa Plus Sim | Simvastatin Alone / Empa Plus Sim / Empa Alone | Empa Plus Sim / Empa Alone / Simvastatin Alone | Empa Plus Sim / Simvastatin Alone / Empa Alone
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (3 Days)
Arm/Group | Empa Alone / Simvastatin Alone / Empa Plus Sim | Empa Alone / Empa Plus Sim / Simvastatin Alone | Simvastatin Alone / Empa Alone / Empa Plus Sim | Simvastatin Alone / Empa Plus Sim / Empa Alone | Empa Plus Sim / Empa Alone / Simvastatin Alone | Empa Plus Sim / Simvastatin Alone / Empa Alone
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (3 Days)
Arm/Group | Empa Alone / Simvastatin Alone / Empa Plus Sim | Empa Alone / Empa Plus Sim / Simvastatin Alone | Simvastatin Alone / Empa Alone / Empa Plus Sim | Simvastatin Alone / Empa Plus Sim / Empa Alone | Empa Plus Sim / Empa Alone / Simvastatin Alone | Empa Plus Sim / Simvastatin Alone / Empa Alone
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 2 | 3 | 3 | 3 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: All subjects who took at least 1 dose of investigational treatment.
Groups:
- Study Overall: This was a randomised, 3-period, crossover trial. The trial was open label. The three treatments were separated by a washout period of at least 7 days.
Arm/Group | Study Overall
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Empa: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 extrapolated to infinity.
  The geometric mean (gMean) and geometric coefficient of variation (gCV) are adjusted values.
Time Frame: 0 hours (h), 20minutes (min), 40min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h after drug administration
Population: Pharmacokinetic (PK) set: PK set included all evaluable subjects who took at least one dose of investigational treatment and provided at least one observation for at least one primary PK endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa Alone: 25mg empagliflozin (empa) alone
- Empa Plus Sim: 25 mg empagliflozin (empa) together with 40 mg simvastatin (sim)
Arm/Group | Empa Alone | Empa Plus Sim
Number analyzed (Participants) | 18 | 18
nmol*h/L | 5571.70 (5.4) | 5685.69 (5.4)
Statistical Analysis 1: Comparison: Empa Alone vs Empa Plus Sim; Considered characteristic is empa plus simvastatin divided by empa alone; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 102.05, 90% CI 2-sided [98.90 to 105.29], Standard Deviation 5.4 — Standard deviation is actually the geometric coefficient of variation (gCV)

2. Primary Outcome: Simvastatin: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity. Simvastatin acid is an active metabolite of simvastatin.
  The geometric mean (gMean) and geometric coefficient of variation (gCV) are adjusted values.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Simvastatin Alone: 40 mg simvastatin alone
Arm/Group | Simvastatin Alone | Empa Plus Sim
Number analyzed (Participants) | 17 | 18
ng*h/mL
  AUC of simvastatin | 33.51 (40.4) | 33.93 (40.4)
  AUC of simvastatin acid | 16.83 (25.5) | 17.65 (25.5)
Statistical Analysis 1: Comparison: Simvastatin Alone vs Empa Plus Sim; AUC of simvastatin Considered characteristic is empa plus simvastatin divided by simvastatin alone; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 101.26, 90% CI 2-sided [80.06 to 128.07], Standard Deviation 40.4 — Standard deviation is actually the gCV
Statistical Analysis 2: Comparison: Simvastatin Alone vs Empa Plus Sim; AUC of simvastatin acid Considered characteristic is empa plus simvastatin divided by simvastatin alone; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 104.87, 90% CI 2-sided [90.09 to 122.07], Standard Deviation 25.5 — Standard deviation is actually the gCV

3. Primary Outcome: Empa: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of the analyte in plasma, per period.
  The geometric mean and geometric coefficient of variation (gCV) are adjusted values
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Alone | Empa Plus Sim
Number analyzed (Participants) | 18 | 18
nmol/L | 774.06 (21.1) | 847.49 (21.1)
Statistical Analysis 1: Comparison: Empa Alone vs Empa Plus Sim; Considered characteristic is empa plus simvastatin divided by empa alone; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 109.49, 90% CI 2-sided [96.91 to 123.69], Standard Deviation 21.1 — Standard deviation is actually the gCV

4. Primary Outcome: Simvastatin: Maximum Measured Concentration (Cmax)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Simvastatin Alone | Empa Plus Sim
Number analyzed (Participants) | 17 | 18
ng/mL
  Cmax of simvastatin | 7.88 (41.7) | 7.65 (41.7)
  Cmax of simvastatin acid | 1.51 (22.7) | 1.47 (22.7)
Statistical Analysis 1: Comparison: Simvastatin Alone vs Empa Plus Sim; Cmax of simvastatin. Considered characteristic is empa plus simvastatin divided by simvastatin alone; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 97.18, 90% CI 2-sided [76.30 to 123.77], Standard Deviation 41.7 — Standard deviation is actually the gCV
Statistical Analysis 2: Comparison: Simvastatin Alone vs Empa Plus Sim; Cmax of simvastatin acid. Considered characteristic is empa plus simvastatin divided by simvastatin alone; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 97.27, 90% CI 2-sided [84.90 to 111.44], Standard Deviation 22.7 — Standard deviation is actually the gCV

5. Secondary Outcome: Empa: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point.
  The geometric mean and geometric coefficient of variation (gCV) are adjusted values.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Alone | Empa Plus Sim
Number analyzed (Participants) | 18 | 18
nmol*h/L | 5481.31 (5.8) | 5619.60 (5.8)
Statistical Analysis 1: Comparison: Empa Alone vs Empa Plus Sim; Considered characteristic is empa plus simvastatin divided by empa alone; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 102.52, 90% CI 2-sided [99.10 to 106.06], Standard Deviation 5.8 — Standard deviation is actually the gCV

6. Secondary Outcome: Simvastatin: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Simvastatin Alone | Empa Plus Sim
Number analyzed (Participants) | 17 | 18
ng*h/mL
  AUC of simvastatin | 31.82 (41.7) | 32.57 (41.7)
  AUC of simvastatin acid | 14.86 (24.8) | 16.53 (24.8)
Statistical Analysis 1: Comparison: Simvastatin Alone vs Empa Plus Sim; AUC of simvastatin. Considered characteristic is empa plus simvastatin divided by simvastatin alone; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 102.34, 90% CI 2-sided [80.39 to 130.29], Standard Deviation 41.7 — Standard deviation is actually the gCV
Statistical Analysis 2: Comparison: Simvastatin Alone vs Empa Plus Sim; AUC of simvastatin acid. Considered characteristic is empa plus simvastatin divided by simvastatin alone; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 111.25, 90% CI 2-sided [95.93 to 129.02], Standard Deviation 24.8 — Standard deviation is actually the gCV

ADVERSE EVENTS:
Time Frame: First administration of trial medication until next administration of trial medication or up to post-study visit, up to 36 days
Arm/Group | Empa Alone | Simvastatin Alone | Empa Plus Sim
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 6/18 | 4/17 | 5/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa Alone (N=18) | Simvastatin Alone (N=17) | Empa Plus Sim (N=18)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0
Purulence (Infections and infestations) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes